CLINICAL TRIAL: NCT00802048
Title: Study of Effectiveness of a Ropivacaïne Continuous Sternal Infusion to Reduce Postoperative Hyperalgesia Induced by Sternotomy After Cardiac Surgery
Brief Title: Local Anesthetic Infusion and Sternotomy
Acronym: CARDIODOLAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUBX2007/26
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Hyperalgesia; Pain
Keywords: Sternotomy; Postoperative hyperalgesia; Intralesional anesthetic infusion; Ropivacaïne; Chronic; Postoperative pain; Cardiac surgery; Sternum; Cardiac surgical procedures
MeSH Terms: conditions — Hyperalgesia; Pain; Bronchiolitis Obliterans Syndrome; Pain, Postoperative | interventions — Anesthetics, Local; Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 48h postoperative infusion of ropivacaine
  Interventions: Drug: Local anesthetic (Ropivacaine)
- 2 (Placebo Comparator): 48h postoperative infusion of NaCl.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Local anesthetic (Ropivacaine) — Local anesthetic infusion
  Arms: 1
Drug: Saline — Saline serum infusion
  Arms: 2

SUMMARY:
Cardiac surgery often induces acute postoperative pain and moreover chronic dysesthesia frequently occur long-term after sternotomy. The high doses of intraoperative opioïds are well known to enhance postoperative hyperalgesia (HA) and a perioperative local anesthetic agent infusion is one of the therapeutic strategies used to limit this phenomena. The aim of this study was to evaluate the effectiveness of a continuous Ropivacaïne sternal infusion compared with a saline serum infusion to limit postoperative HA, pain and morphine consumption (M) after sternotomy in cardiac surgery.

This strategy could lead to lower postoperative morphine consumption and opioïd induced hyperalgesia.

DETAILED DESCRIPTION:
* Principal Objective: comparison of peri-incisionnal dynamic hyperalgesia extend evaluated by Von Frey filament during the first postoperative week between the two groups.
* Secondary Objective: comparison of peri-incisionnal static hyperalgesia (pain threshold) extend evaluated by Von Frey filament, postoperative pain scores, morphine consumption, hemodynamic and respiratory parameters during the first postoperative week and incidence of chronic pain and dysesthesia at six month between the two groups. Ropivacaïne plasmatic concentration will be monitored, during infusion.
* Study design : monocentric, double blind randomized clinical trial comparing two groups of patients with a same intraoperative anesthetic management :

  * Group 1: Ropivacaïne infiltration before skin incision followed by a 48 hours Ropivacaïne continuous infusion after surgery through a sternal fenestrated catheter
  * Group 2: same protocol with pre and postoperative saline infusion

Postoperative pain management is identical in the two groups based upon a Morphine sulfate PCA pump for the first 48 hours.

• Number of subjects : 40 patients, 20 in each group

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 50 to 75 years old
* ASA score : 1-3
* Cardiac surgery with median sternotomy for:

  * single valve replacement, Bentall, Bahnson, Tyrone David procedure
  * single or multiple Cardiac Artery Bypass Grafting (CABG)
  * combined surgery (valve replacement + CABG)
  * without predicted risk of postoperative complication
* Informed consent obtained from the patient
* Patient beneficiating of social insurance

Exclusion Criteria:

* patient refusal to participate in the study
* Drug or alcohol abuse history
* Analgesic or opioid consumption within the 12 hours preceding the surgery
* Chronic use of analgesic drugs or history of chronic pain
* Disability to understand morphine PCA use
* Allergy to ropivacaine or other local anaesthesia
* Patient treated by fluvoxamine or enoxamine
* Patient suffering for liver insufficiency (child score >A)
* Patient with major preoperative hypovolemia

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
hyperalgesia area size around the cicatrix | 24h after surgery

SECONDARY OUTCOMES:
Peroperative monitoring datas | Peroperative
Dynamic hyperalgesia | Day 2, 3 and 6
Static hyperalgesia | Day 1, 2, 3 and 6
Ropivacaine plasmatic concentration | 24h and 48h

CONTACTS AND LOCATIONS:
Overall Officials: Olivier POUQUET, Dr, Principal Investigator — University Hospital, Bordeaux; Antoine BENARD, Dr, Study Chair — University Hospital, Bordeaux; Mathieu LAFARGUE, MD, Principal Investigator — University Hospital, Bordeaux; Alexandre OUATTARA, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Département d'Anesthésie-Réanimation II - Hôpital cardiologique - Groupe Hospitalier Sud, CHU de Bordeaux - 4, Av de Magellan, Pessac, France